CLINICAL TRIAL: NCT07099170
Title: Comparison of Training Models in Pelvic Floor Muscle Training in Healthy Adult Women
Brief Title: Training Models in Pelvic Floor Muscle Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ipek Yavas, PT, MSc, Lecturer, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IzmirUEcon-PTR-01
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Muscle Exercise; Healthy Adult Women; Pelvic Floor Muscle Training
Keywords: pelvic floor muscle training; pelvic floor muscle exercise; Healthy Adult Women; Comparison Models

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brochure-Based Pelvic Floor Muscle Training (Experimental)
  Interventions: Behavioral: Brochure-Based Pelvic Floor Muscle Training
- Verbal Instruction-Based Pelvic Floor Muscle Training (Experimental)
  Interventions: Behavioral: Verbal Instruction-Based Pelvic Floor Muscle Training
- Visual-Aided Pelvic Floor Muscle Training (Experimental)
  Interventions: Behavioral: Visual-Aided Pelvic Floor Muscle Training
- External Palpation-Aided Pelvic Floor Muscle Training (Experimental)
  Interventions: Behavioral: External Palpation-Aided Pelvic Floor Muscle Training

INTERVENTIONS:
Behavioral: Brochure-Based Pelvic Floor Muscle Training — Brochure-based pelvic floor muscle training will be conducted by providing participants with a brochure containing information about the anatomy, functions, and importance of the pelvic floor, as well as instructions on how to contract the pelvic floor muscles. All educational content will be delivered solely through the brochure, and no additional verbal or written information will be provided to the participants. The brochure will include detailed explanations of pelvic floor muscle contractions and imagery techniques. Participants will be given 30 minutes to review the brochure and apply the training independently.
  Arms: Brochure-Based Pelvic Floor Muscle Training
Behavioral: Verbal Instruction-Based Pelvic Floor Muscle Training — Verbal instruction-based pelvic floor muscle training involves providing participants with information about the anatomy, functions, and importance of the pelvic floor, as well as instruction on how to correctly contract the pelvic floor muscles. All explanations will be delivered verbally, and no additional equipment or visual aids will be used. During the training, imagery techniques based on verbal cues will be employed. Commonly used metaphors such as a hammock, a faucet, an elevator, or a ship will be utilized to facilitate imagery. Participants will be asked to focus on their pelvic floor and imagine the contractions, and they will be informed about the potential effects of these contractions during the session.
  Arms: Verbal Instruction-Based Pelvic Floor Muscle Training
Behavioral: Visual-Aided Pelvic Floor Muscle Training — Visual-aided pelvic floor muscle training includes providing participants with information about the anatomy, functions, and importance of the pelvic floor, as well as training on how to properly contract the pelvic floor muscles. The training will be conducted using anatomical models, visual materials, and videos. Following the explanation of pelvic floor anatomy with models and visual aids, the function and importance of the pelvic floor will be presented through video demonstrations. During the session, the pelvic floor will be visually represented using common metaphors such as a hammock, a faucet, an elevator, or a ship, and these visuals will support the use of imagery techniques. Participants will be asked to focus on their pelvic floor and imagine the contractions, and they will be provided with information about the expected effects of the contractions.
  Arms: Visual-Aided Pelvic Floor Muscle Training
Behavioral: External Palpation-Aided Pelvic Floor Muscle Training — External Palpation-Aided Pelvic Floor Muscle Training This training involves educating participants on the pelvic floor's anatomy, function, and importance, along with instructions on proper muscle contraction. After an educational session using anatomical models, visuals, and videos, external palpation is used to guide correct muscle activation. In a hook-lying position and fully clothed, participants receive light, transverse pressure from a physiotherapist on key pelvic floor muscles (ischiocavernosus, bulbospongiosus/bulbocavernosus, or perineum). The therapist observes real-time muscle response, provides feedback, and offers verbal cues. Imagery techniques (e.g., hammock, faucet, elevator, ship) may be used to support motor learning and awareness.
  Arms: External Palpation-Aided Pelvic Floor Muscle Training

SUMMARY:
Pelvic floor muscle training (PFMT) is an exercise approach designed to improve the strength, endurance, power, relaxation, or coordination of the pelvic floor muscles. It is recommended as a first-line treatment for urinary incontinence (stress, urge, mixed), pelvic organ prolapse, and fecal incontinence. Evidence also suggests its potential to enhance sexual function in both men and women.

To teach proper pelvic floor contraction, individuals must first learn the anatomical location, structure, and function of these muscles. Various teaching strategies can support motor learning, such as verbal cues (commands or imagery), visual input (anatomical models or illustrations), physical guidance (tactile feedback), and environmental adjustments (comfortable positions, safe space). Yet, the choice of teaching method in clinical practice is currently based only on experience, not evidence.

This study aims to compare the effectiveness of four different PFMT teaching models-brochure-based, verbal instruction-based, visual instruction-based, and external palpation-aided-in teaching correct pelvic floor contraction and improving awareness in healthy adult women. It will be conducted as a four-arm randomized controlled trial. Participants will be evaluated before the training, immediately after, and one week later.

The findings from this study will help identify the most effective and practical approach for teaching PFMT. Although the study is conducted with healthy women without pelvic symptoms, the results will inform better training strategies for individuals with pelvic floor dysfunction, including those with urinary problems, chronic diseases, or pregnancy-related pelvic floor issues. Ultimately, this research seeks to fill a gap in the current literature and contribute to more evidence-based clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Female
* Willingness to participate in the study

Exclusion Criteria:

* Pregnancy
* History of cesarean or vaginal delivery within the past 6 months
* Previous pelvic floor muscle training
* History of pelvic surgery
* Currently receiving or having received treatment for pelvic organ prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
Mean Bladder Base Displacement During Pelvic Floor Muscle Contraction | Baseline (pre-training), immediately after training (within 1 hours of completion of training), and follow-up (7 days after training)
  Pelvic floor muscle activity will be objectively assessed using transabdominal B-mode ultrasound, which allows real-time visualization of muscle movement.
  Participants will drink 500 ml of water and refrain from voiding before the test. While lying supine with knees flexed, a linear probe will be placed transabdominal suprapubically to visualize the bladder base. Bladder displacement during pelvic floor contraction will be measured by placing markers on the ultrasound image at rest and during contraction. The procedure will be repeated three times, and the average measurement in millimeters will be recorded.
Presence or Absence of Voluntary Pelvic Floor Muscle Contraction Assessed by Palpation | Baseline (pre-training), immediately after training (within 1 hours of completion of training), and follow-up (7 days after training)
  The participants' ability to contract their pelvic floor muscles will be assessed by a specialized physiotherapist through external palpation and categorized as no voluntary contraction, weak, moderate, or strong contraction.

SECONDARY OUTCOMES:
Semi-Structured Form for Pelvic Floor Awareness | Baseline (pre-training), immediately after training (within 1 hours of completion of training), and follow-up (7 days after training)
  A semi-structured questionnaire was developed to assess participants' knowledge and awareness regarding pelvic floor anatomy, function, dysfunction, and exercises.
Participant Satisfaction | Immediately after training (within 1 hours of completion of training)
  Participant satisfaction with the training program will be assessed immediately after the intervention using a Visual Analog Scale (VAS). Participants will be asked to respond to two questions: (1) "How satisfied are you with the training you received?" and (2) "Do you think the training you received was useful?" Each question will be rated on a scale from 0 to 10, where 0 indicates "Not satisfied at all" or "Not useful at all" and 10 indicates "Extremely satisfied" or "Extremely useful." The responses will be recorded as continuous variables.

OTHER OUTCOMES:
Sociodemographic and Clinical Information | Baseline (pre-training)
  Data on age, sex, smoking status, employment status, marital status, regular exercise habits, and medical history will be collected using the form provided in the appendix.
Anthropometric | Baseline (pre-training)
  body weight.
Anthropometric - height | Baseline (pre-training)
  height
Kinesthetic and Visual Imagery Questionnaire | Baseline (pre-training)
  Questionnaire evaluates participants' ability to visualize (visual imagery) and feel (kinesthetic imagery) the movements. It consists of 10 movements.
  For each item, participants first perform the movement, then imagine watching themselves perform it and rate the clarity of the image on a 5-point scale (1 = no image, 5 = as clear as real). Next, they repeat the movement and then imagine performing it, focusing on the sensation, and rate the intensity (1 = no sensation, 5 = as intense as real). This process is repeated for all 10 movements.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir University of Economics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No